CLINICAL TRIAL: NCT04075695
Title: Ultra-wide-field Fluorescein Angiography in Patients With Retinal Vein Occlusion
Acronym: UWFARVO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Changzheng Chen, Chief of Department of Ophthalmology, Renmin Hospital of Wuhan University
Other Study IDs: UWFARVO
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Retinal Vein Occlusion
Keywords: ischemic index; Ultra-wide field fundus fluorescein angiography; vascular leakage index
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The changes of ischemic index and vascular leakage index, and the effect on macular edema and neovascularization in retinal vein occlusion by ultra-wide field fluorescence angiography (UWFA)

DETAILED DESCRIPTION:
In this study, the ischemic index and vascular leakage index, and the effect on macular edema and neovascularization in retinal vein occlusion will be evaluated by ultra-wide field fluorescence angiography (UWFA). UWFA has a wider range than conventional angiography, and can clearly observe the peripheral retina. The purpose of this study is to quantitatively analyze these changes and investigate the effect on macular edema and neovascularization secondary to retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or more
2. Patients with a diagnosis of CRVO,BRVO or HRVO without macular edema
3. Duration of RVO not more than 4 months
4. Naïve patients. Patient with previous RVO (more than 12 months before the inclusion date) which completely resolved (normalization of visual acuity and fundus examination) and who experienced a recurrence of RVO are also considered naive
5. Patient who agrees to participate to the study and who has given his/her written, informed consent

Exclusion Criteria:

1. Patient with another retinal disease in the study eye: diabetic retinopathy, maculopathy of any cause (age-related macular degeneration, epimacular membrane, myopia, etc) responsible for decreased vision, advanced glaucoma, cataract severely affecting vision and/or requiring surgical treatment during the 24 months study period
2. Active or suspected ocular or periocular infection
3. Active severe intraocular inflammation
4. RVO complicated with neovascularization
5. Patient who has previously undergone laser panretinal photocoagulation, grid-laser or photodynamic therapy, any anti-VEGF or corticoids intravitreal injections in the study eye
6. Patient already included in the study for the treatment of the fellow eye
7. Pregnant or breastfeeding woman
8. Lack of effective contraception for women of childbearing age
9. Patient taking part in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Change in non-perfused areas in different retinal area | Baseline and1，2，3，6，9and 12 months
  Change in non-perfused areas in different retinal area from Baseline to 1，2，3，6，9and 12 months

SECONDARY OUTCOMES:
Change in best corrected visual acuity | Baseline and1，2， 3, 6, 9 and 12 months
  Change in best corrected visual acuity from Baseline to 1，2，3，6，9and 12 months
Change in central macular thickness | Baseline and1，2， 3, 6, 9 and 12 months
  Change in central macular thickness from Baseline to 1，2，3，6，9and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renmin Hospital of Wuhan University, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China